CLINICAL TRIAL: NCT05116878
Title: Enhancing Facial Nerve Neuroprotection and Regeneration Through Omega-3 Supplementation Following Vestibular Schwannoma Resection
Brief Title: Enhancing Facial Nerve Function With Omega-3 After Resection of Vestibular Schwannoma
Acronym: EFFORTS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Funding.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael J. Link, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-007120
Record Dates: First submitted 2021-11-02; First posted 2021-11-11 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Vestibular Schwannoma
Keywords: Facial nerve outcomes; Vestibular schwannoma resection; Acoustic neuroma; Omega-3; Nerve regeneration; Neuroprotection
MeSH Terms: conditions — Neuroma, Acoustic | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All patients and clinical providers, including outcomes assessors, will be blinded to treatment vs placebo arms. Masking will be performed by an independent trial coordinator not involved with data collection, data analysis, or patient care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Omega-3 Group (Experimental): Subjects will receive omega-3 supplementation (Nature's Bounty Fish Oil 1400 mg, containing 980 mg Omega-3 per capsule), to begin taking 3 days prior to surgical resection of their vestibular schwannoma. Subjects will continue to take the omega-3 supplementation for 6 weeks post-operatively.
  Interventions: Dietary Supplement: Omega-3
- Placebo Group (Placebo Comparator): Subjects will receive a placebo to begin taking 3 days prior to clinical care of surgical resection of vestibular schwannoma. Subjects will continue to take the placebo for 6 weeks post-operatively.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 — One capsule orally twice daily beginning 3 days prior to clinical care surgical intervention and continuing 6 weeks post-operative
  Arms: Omega-3 Group
Dietary Supplement: Placebo — One cellulose capsule orally twice daily beginning 3 days prior to clinical care surgical intervention and continuing 6 weeks post-operative
  Arms: Placebo Group

SUMMARY:
The purpose of this research is to develop a therapeutic agent to help improve facial nerve outcomes and ultimately improve long-term quality-of-life following surgical resection of vestibular schwannomas. It is possible the therapeutic agent may impact tumor control rates as well, and this will also be studied. Using rigorous scientific methods, we will assess whether these factors are impacted by the treatment agent (Omega-3) versus placebo control (cellulose).

DETAILED DESCRIPTION:
Vestibular schwannomas (VS) are common, often-benign intracranial neoplasms, however surgical resection carries high risk of causing neurologic impairments that may severely impact patient quality-of-life. The most morbid common postoperative deficit is facial weakness due to the close anatomic proximity of VS with the facial nerve, which is frequently stretched and attenuated by the tumor itself, and subject to additional mechanical stress during surgery. In addition to disfiguring cosmesis, facial weakness carries the secondary effects of abnormal speech, ocular morbidity from inadequate eye closure and corneal lubrication, and dysfunctional swallowing mechanics. Some patients may eventually recover partial facial nerve function; however, this is an unreliable process that proceeds slowly over months to years, if at all. At present, no pharmacologic avenue exists for promoting facial nerve neuroprotection or regeneration. Correspondingly, the development of a therapeutic agent to stimulate improved facial nerve outcomes would markedly enhance patient outcomes and quality-of-life.

In the anterior skull base, loss of olfaction is a common sequela of following endoscopic surgical resection due to direct nerve manipulation, impacting approximately 25% of patients who undergo endoscopic endonasal tumor resection. In a recent randomized clinical trial, postoperative supplementation with omega-3 yielded a significant, sustained 1-2-point improvements on the University of Pennsylvania Smell Identification Test as assessed at six weeks, three months, and six months post-operatively. Although mechanistic understanding of the relationship between omega-3 supplementation and olfactory function preservation is incompletely understood, preliminary data support the hypothesis of direct neural regeneration and/or neuro-protective effects through anti-demyelination effects. More specifically, polyunsaturated fatty acids have been shown to modulate neural plasticity and provide a protective role in maintaining functional neuronal cell membranes thought to be critical for maintaining nerve connectivity and function. It is also possible that omega-3, a known anti-inflammatory agent through reducing local IL-6, TNF, NFkB, impacts the innate immune system to mitigate demyelination and other destructive post-treatment inflammatory injuries to cranial nerves and surrounding support cells. Given the highly interrelated mechanisms-of-injury resulting in olfactory deficit after anterior skull base surgery and facial weakness after VS resection, application of omega-3 fatty acids may provide similar benefits with respect to facial nerve protection and/or rehabilitation. As a fascinating aside, new pre-clinic animal model evidence also suggests that omega-3 fatty acid supplementation may result in delayed progression in a neuroblastoma xenograft model. These effects are attributed to anti-inflammatory and anti-angiogenic effects via anti-VEGF and other anti-proliferative growth factors; factors also implicated in VS pathophysiology, suggesting that omega-3 may also impact early tumor control as well. We hypothesize that post-operative omega-3 supplementation will improve facial nerve function following resection of vestibular schwannomas and enhance early tumor control rates.

ELIGIBILITY:
Inclusion Criteria:

* VS on final pathology report
* Surgical intervention (RS, MF, TL, other)
* Primary and revision cases included, including prior radiation

Exclusion Criteria:

* History of liver disease or abnormal liver function tests
* Diabetic patients with specific contraindication to omega-3 supplementation
* History of bleeding disorder, or recommended use of anticoagulation (not including anti-platelets or NSAIDs) during the treatment period
* Neurofibromatosis 1 or 2, or schwanomatosis disorders
* Non-VS pathology
* Patients already taking fish oil/omega-3 supplementation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
Change in facial nerve function | Baseline, 3 and 12 months post-operative
  Subjects will receive independent examination by at least three expert clinical assessors using the standardized, and clinically validated, House-Brackmann facial function score to characterize the severity of facial paralysis. Score is determined by measurements (in cm) of subjects movements of facial reference points on a scale of 0-8 which translate to grading system of grade I (normal) - Grade VI (no facial motion)
Tumor Control | 12 months post-operative
  Number of subjects to have tumor recurrence or progression of vestibular schwannoma as assessed by post-operative radiography (MRI) imaging

CONTACTS AND LOCATIONS:
Overall Officials: Michael Link, MD, Principal Investigator — Mayo Clinic; Lucas P Carlstrom, MD, PhD, Study Director — Mayo Clinic; Matthew L Carlson, MD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
May be available on specific requests for collaboration.

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials